CLINICAL TRIAL: NCT01565785
Title: Self-Management Guided Discharge Teaching for Parents of Hospitalized Children: A Pilot Study
Brief Title: Evaluating a New Way to Prepare Parents of Hospitalized Children for Discharge and Management of Child at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); University of Wisconsin, Milwaukee (Other); Marquette University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 259192-1
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Patient Discharge
Keywords: Child parent home self-management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Discharge Prepartion with The FSM-DPI (Experimental): 25 families on each of 2 units will receive the will receive the Family Self-Management-Discharge Preparation Intervention (FSM-DPI). This scripted theory-based intervention is delivered by the study nurse using a e-mobile device. Eight elements of discharge preparation are addressed, the nurse assesses the family status and documents the additional care provided.
  Interventions: Behavioral: The FSM-DPI.
- control group (No Intervention): 25 parents on each unit receiving standard of care in discharge preparation.

INTERVENTIONS:
Behavioral: The FSM-DPI. — Nurses will assess key elements of family self-management (home care, child's care, practice, medications, watching child, recovery, development, family adjustment and parental support) and address any deficits to facilitate effective discharge and family management of child at home after hospitalization.
  Other Names: Tailored; behavioral
  Arms: Discharge Prepartion with The FSM-DPI

SUMMARY:
The purpose of this study is to pilot test the 'Family Self- Management Discharge Preparation Intervention [FSM-DPI]' that focuses on content and delivery methods to support an effective family transition to home self-management after a child's hospitalization.

DETAILED DESCRIPTION:
The specific aims of the study are:

1. To estimate the effect of an intervention designed to improve family self-management after discharge of a hospitalized child on:

   1. Family self-management process (e.g., knowledge, self-regulation, and social facilitation)
   2. Proximal family self-management behavioral outcomes, (e.g., post-discharge parental coping difficulty and family impact), and unplanned use of post-discharge services (calls to family/friends, health care providers, hospital; unscheduled office visits, urgent care/ED visits, readmission).
2. To describe nurse assessment and patient responses to the FSM-DPI.
3. To compare nurse satisfaction with discharge teaching process when nurses perform discharge teaching using the FSM-DPI vs. the standard discharge teaching approach.

A novel discharge preparation intervention delivered by nurses to parents of hospitalized children who are being discharged home was developed based on previous research conducted by the investigators. The intervention is grounded in the individual and family self-management Theory. To test the impact of the intervention on discharge preparation process and parent outcomes, the investigators will conduct a pilot trial implementation using trained staff nurses to deliver the intervention. To measure the effects of the intervention a difference- in-differences approach with be used with selection of 200 parents with 50 in each of 4 groups: Baseline control 1 (parents assigned for usual care to study nurses before training on the use of the intervention); Baseline control group 2 ( parent assigned for usual care to other than study nurses); Implementation group ( parents assigned to study nurses who will receive the intervention); Concurrent control group ( parent assigned to other than study nurses). The study will be conducted on two nursing units and half of the sample will be selected from each unit using a random selection procedure.

Data to be collected from all parents (baseline control, implementation, concurrent control) on the day of hospital discharge include: Parent enrollment sheet for collection of parent demographics; Quality of Discharge Teaching Scale, Readiness for Hospital Discharge Scale, Care Transition Measure. In addition the CHW Synergy form will be copied from the child's medical record to provide information on child characteristics of the hospitalization. At 3 weeks post-discharge, parents will be contacted by telephone to obtain outcome data using the Post-Coping Difficulty Scale and the PedsQL™. Parents will also be asked questions about post-discharge utilization of health services.

Nurses will record process measures related to the delivery of the intervention. In addition the nurse of parents in implementation and control groups will complete assessments of patient readiness for discharge using the Readiness for Hospital Discharge Scale and will rate their experience with the discharge process on a survey developed by the research team.

Analysis will provide information about the utility of the FSM-DPI and preliminary data on which to base revisions and enhancements to the intervention and for development of a larger implementation trial.

ELIGIBILITY:
Inclusion Criteria:

* Parents must be at least 18 years of age, speak sufficient English to complete paper or online questionnaires, have a child who has been in the hospital for 2 days and is expected to go home on the data of data collection

Exclusion Criteria:

* Parents will be excluded if their child is discharged home to hospice care, or if they were in the hospital less than 2 days, were admitted as a short stay, or remain in the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Post-Coping Difficulty | 3 weeks after discharge
  The Post-Coping Difficulty Scale is a measure of parent perception of difficulty and ability to manage their child's care at home.

SECONDARY OUTCOMES:
Pediatric Quality of Life (parent report) | 3 weeks after discharge
  The child quality of life (parent as reporter) is a measure with total score and 4 domain scores, physical, emotional, social and school.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen J Sawin, PhD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin; Marianne Weiss, DNSc, RN, Principal Investigator — Marquette University
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States